CLINICAL TRIAL: NCT05764772
Title: Validation of Photon Counting/Spectral Computed Tomography Angiography of Carotid Plaque Composition in Patients With Ischemic Stroke
Brief Title: CT Evaluation of Carotid Plaque Components
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jae W. Song, MD, MS, Principal Investigator, University of Pennsylvania
Other Study IDs: 852646
Record Dates: First submitted 2023-02-10; First posted 2023-03-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Carotid Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to validate the diagnostic performance of photon counting/spectral CT to distinguish tissue components in ischemic stroke with MRI, semi-automated segmentation software or histology as the reference standard.

The main question[s] it aims to answer are:

1. Presence or absence of calcium, hemorrhage, and lipid plaque components as determined on CT will be confirmed with carotid MRI, segmentation quantitative (e.g., volume) output from segmentation software, or histologic staining.
2. Volumes of hemorrhage, lipid, and calcium components will be measured to determine plaque phenotype and correlated with ipsilateral intracranial stroke burden.

Participants will be asked to do the following:

Aim 1:

* 1 Photon counting/spectral CT angiography of the neck
* 1 Research Carotid/Neck MRI of the carotid arteries (if eligible)

Aim 2:

* 1 Research Carotid/Neck MRI of the carotid arteries (if eligible)
* 1 Photon counting/spectral CT angiography of the neck
* 1 Carotid plaque tissue from participants surgery will be retrieved, imaged, and stained (if eligible)

DETAILED DESCRIPTION:
Independent of the degree of stenosis, specific features of carotid plaque composition are associated with a high risk of thromboembolic and recurrent stroke. Many lines of evidence show a significant association between the presence of intraplaque hemorrhage and lipid rich necrotic core in carotid plaque independent of vessel stenosis in patients with ipsilateral ischemic infarcts. In fact, up to 17% of ischemic strokes are classified as embolic stroke of undetermined source (ESUS) after a comprehensive diagnostic work-up. A subset of these patients have stroke due to mildly stenotic plaque composed of high-risk non-calcified carotid plaque components that are presently difficult to distinguish by noninvasive conventional imaging tests. Presently first-line imaging of acute stroke patients is computed tomography angiography (CTA) of the head and neck. Although conventional CTA provides information about stenosis, it lacks the ability to distinguish tissue components with similar attenuation curves (e.g., lipid and intraplaque hemorrhage). Thus, invaluable diagnostic information is lost due to limitations of conventional CTA. By contrast, photon-counting/spectral CT is a novel technology that can identify material-specific characteristics and identify plaque components (e.g., iron/hemorrhage, lipid, and calcium) based on the specific behavior of these materials at different photon energy levels.

The investigators propose testing the diagnostic performance of this new CT technology to detect different plaque components in subjects who are medically managed by carotid MRI or postprocessing PCCT images using a semi-automated carotid plaque segmentation software. The investigators also propose testing the diagnostic performance of this new CT technology in patients undergoing carotid endarterectomy revascularization surgery as standard of care with carotid MRI and histologic validation of the resected plaque tissue (ground truth).

Accurate detection of these high-risk noncalcified plaque components by noninvasive imaging methods would be of great value to identifying a patient population at highest risk for embolic stroke from carotid disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic carotid stenosis with ipsilateral ischemic infarcts attributable to the carotid disease
* At least 1mm of noncalcified plaque on same side of stroke
* Brain MRI documenting ischemic infarct in distribution attributable to ipsilateral carotid disease
* Patients planned to undergo carotid endarterectomies
* Patients must be able to read and understand English
* Participants must sign the informed consent form

Exclusion Criteria:

* Exclusion Criteria

  * Patients less than 18 years old
  * Women who are pregnant and/or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute stroke or transient ischemic attacks and stenosis of the ipsilateral carotid artery will be identified and eligible patients will be screened and consented for study participation in a multi-disciplinary effort by Vascular Neurology (contact: Dr. Brett Cucchiara), Vascular Surgery (contact: Dr. Grace Wang), and Diagnostic Radiology (contact: Dr. Jae W. Song).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To validate the diagnostic performance of photon counting/spectral CT | 3years
  Presence or absence of calcium, hemorrhage, and lipid plaque components as determined on CT will be confirmed with carotid MRI, segmentation quantitative (e.g., volume) output from segmentation software, or histologic staining.

CONTACTS AND LOCATIONS:
Overall Officials: Jae W Song, Principal Investigator — University of Pennsylvania Hospital
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States